CLINICAL TRIAL: NCT03674749
Title: Effect of Meditation and Hyperbaric Oxygen Therapy on Cognition, Healing Process and Overall Well-being in Elderly Patients With Chronic Wounds
Brief Title: The Effects of Meditation and Hyperbaric Oxygen Therapy on Chronic Wounds
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18-5271
Record Dates: First submitted 2018-09-14; First posted 2018-09-18 (Actual); Last update posted 2019-12-16 (Actual); Status verified 2019-12

CONDITIONS: Wound
MeSH Terms: conditions — Wounds and Injuries | interventions — Meditation

STUDY DESIGN:
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hyperbaric Oxygen (Active Comparator): Hyperbaric oxygen treatment with 100% oxygen at 2.0 ATA for 90 min, once daily, five times a week for 8 consecutive weeks
  Interventions: Other: Meditation and Hyperbaric Oxygen Treament
- Meditation with Hyperbaric Oxygen (Experimental): Meditation session combined with each hyperbaric oxygen treatment with 100% oxygen at 2.0 ATA for 90 min, once daily, five times a week for 8 consecutive weeks,
  Interventions: Other: Meditation and Hyperbaric Oxygen Treament

INTERVENTIONS:
Other: Meditation and Hyperbaric Oxygen Treament — Meditation sessions will be combined with hyperbaric oxygen treatment

SUMMARY:
In Ontario, wound care support has steadily increased over the years. With the growth of the aging population, the financial and psychological burden related to wound care will continue to rise. Studies have shown that structured meditation programs can improve on the recovery process for both physical and psychological disease. Therapeutic treatments like Hyperbaric Oxygen Therapy (HBOT) for chronic wounds have shown to promote angiogenesis, cerebral blood and neuroplasticity in patients with stroke, traumatic brain injury and chronic pain. By combining meditation and HBOT, this have been independently shown to improve healing and reducing costs associated with chronic wounds.

DETAILED DESCRIPTION:
Each year, Community Care Access Centers (CCAC) provide long-term wound care for over 22,000 patients in Ontario, with numbers steadily increasing with the aging population. In Ontario, the cost of community care for lower leg ulcers has been estimated at over $500 million per year. This does not include the additional cost of adjunctive HBOT, which averages over $120 thousand for a standard 40 treatment course. These costs are further compounded by the psychological comorbidities that often accompany chronic disease, although these numbers are difficult to capture. Across Canada, the health burden cost of anxiety and depression alone totals over $14 billion annually, with disability costs comparable to those associated with heart disease. Furthermore, recent evidence suggests that psychological interventions are more cost-effective than drug treatment, with comparable results.

The elderly patients with chronic non-healing wounds experience a sense of powerlessness and loss of autonomy that profoundly impacts subjective wellbeing. These psychological effects in turn compromise healing, as growing evidence suggests that psychological stress impacts wound repair [1, 2]. Recent studies have shown that structured meditation programs can improve recovery from both physical and psychological disease. For example, meditation enhances immune response [3, 4] while reducing blood pressure [5], insulin resistance [6], oxidative stress [7], inflammation [8], and other risk indices. Furthermore, meditation therapy can be broadly applied with few limitations, having successfully been used in elderly [9], ill [10] and disabled [11] populations.

Hyperbaric oxygen therapy (HBOT) is an adjuvant therapy for chronic wounds. HBOT increases oxygen delivery to tissues via inhalation of 100% oxygen at high barometric pressures. HBOT has been shown to promote angiogenesis, cerebral blood and neuroplasticity in patients with stroke, traumatic brain injury and chronic pain. Furthermore, HBOT also alleviates inflammation, reduces oxidative stress, inhibits apoptosis and stimulates signaling pathways essential for wound healing.

Patients referred for HBOT assessment often have "problem wounds" that have failed prolonged courses of standard wound care. These refractory wounds may benefit from a multimodal approach that targets both the physical and psychological manifestations of chronic disease. Meditation is a simple and economical addition to HBOT that may further enhance the rate of healing by alleviating psychological stressors. Meditation encompasses a spectrum of mindfulness-based interventions that have been shown to improve mental and physical health in randomized trials. Meditation reduces stress, pain, anxiety, depression and blood pressure while improving cognition and memory performance. A variety of specialties have begun to use meditation as a cost-effective, low-stigma adjunct to standard medical and psychiatric care.

Meditation and HBOT have been independently shown to improve healing, and may have synergistic effects when applied together. This combined intervention has the potential to improve mood while enhancing the healing process, offering improved health while reducing the costs associated with chronic wounds.

ELIGIBILITY:
Inclusion criteria:

1. at least 3 month history of non-healing wounds, affecting lower extremities
2. 55 years

Exclusion criteria:

1. claustrophobia
2. seizure disorder
3. active asthma
4. severe chronic obstructive pulmonary disease
5. history of pneumothorax
6. history of severe congestive heart failure with left ventricular ejection fraction < 25%
7. unstable angina
8. chronic or acute otitis media or major ear drum trauma
9. current treatment with bleomycin, cisplatin, doxorubicin and disulfiram
10. recent relapse of depression, psychosis, schizophrenia, hallucinations, suicidal thoughts

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-09-10 (Actual); Primary Completion 2020-03-31 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of patients finishing the study protocol. | 1 year

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Rouge Valley Medical Centre, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario

REFERENCES:
- [Background] Broadbent E, Petrie KJ, Alley PG, Booth RJ. Psychological stress impairs early wound repair following surgery. Psychosom Med. 2003 Sep-Oct;65(5):865-9. doi: 10.1097/01.psy.0000088589.92699.30. PMID 14508033
- [Background] Gouin JP, Kiecolt-Glaser JK. The impact of psychological stress on wound healing: methods and mechanisms. Immunol Allergy Clin North Am. 2011 Feb;31(1):81-93. doi: 10.1016/j.iac.2010.09.010. PMID 21094925
- [Background] Davidson RJ, Kabat-Zinn J, Schumacher J, Rosenkranz M, Muller D, Santorelli SF, Urbanowski F, Harrington A, Bonus K, Sheridan JF. Alterations in brain and immune function produced by mindfulness meditation. Psychosom Med. 2003 Jul-Aug;65(4):564-70. doi: 10.1097/01.psy.0000077505.67574.e3. PMID 12883106
- [Background] Pace TW, Negi LT, Adame DD, Cole SP, Sivilli TI, Brown TD, Issa MJ, Raison CL. Effect of compassion meditation on neuroendocrine, innate immune and behavioral responses to psychosocial stress. Psychoneuroendocrinology. 2009 Jan;34(1):87-98. doi: 10.1016/j.psyneuen.2008.08.011. Epub 2008 Oct 4. PMID 18835662
- [Background] Goldstein CM, Josephson R, Xie S, Hughes JW. Current perspectives on the use of meditation to reduce blood pressure. Int J Hypertens. 2012;2012:578397. doi: 10.1155/2012/578397. Epub 2012 Mar 5. PMID 22518287
- [Background] Paul-Labrador M, Polk D, Dwyer JH, Velasquez I, Nidich S, Rainforth M, Schneider R, Merz CN. Effects of a randomized controlled trial of transcendental meditation on components of the metabolic syndrome in subjects with coronary heart disease. Arch Intern Med. 2006 Jun 12;166(11):1218-24. doi: 10.1001/archinte.166.11.1218. PMID 16772250
- [Background] Mahagita C. Roles of meditation on alleviation of oxidative stress and improvement of antioxidant system. J Med Assoc Thai. 2010 Nov;93 Suppl 6:S242-54. PMID 21280542
- [Background] Buric I, Farias M, Jong J, Mee C, Brazil IA. What Is the Molecular Signature of Mind-Body Interventions? A Systematic Review of Gene Expression Changes Induced by Meditation and Related Practices. Front Immunol. 2017 Jun 16;8:670. doi: 10.3389/fimmu.2017.00670. eCollection 2017. PMID 28670311
- [Background] Gard T, Holzel BK, Lazar SW. The potential effects of meditation on age-related cognitive decline: a systematic review. Ann N Y Acad Sci. 2014 Jan;1307:89-103. doi: 10.1111/nyas.12348. PMID 24571182
- [Background] Bonadonna R. Meditation's impact on chronic illness. Holist Nurs Pract. 2003 Nov-Dec;17(6):309-19. doi: 10.1097/00004650-200311000-00006. PMID 14650573
- [Background] Squier S. Meditation, disability, and identity. Lit Med. 2004 Spring;23(1):23-45; discussion 61-5. doi: 10.1353/lm.2004.0012. No abstract available. PMID 15264508
- [Background] Harris C, Bates-Jensen B. et al. ,The Bates-Jensen Wound Assessment Tool (BWAT): Development of a Pictorial Guide for Training Nurses. Wound Care Canada, 2009, 7 (2): p 33-38
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Scarpina F, Tagini S. The Stroop Color and Word Test. Front Psychol. 2017 Apr 12;8:557. doi: 10.3389/fpsyg.2017.00557. eCollection 2017. PMID 28446889
- [Background] Geisser ME, Clauw DJ, Strand V, Gendreau MR, Palmer R, Williams DA. Contributions of change in clinical status parameters to Patient Global Impression of Change (PGIC) scores among persons with fibromyalgia treated with milnacipran. Pain. 2010 May;149(2):373-378. doi: 10.1016/j.pain.2010.02.043. Epub 2010 Mar 23. PMID 20332060
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820